CLINICAL TRIAL: NCT02490618
Title: The Use of a Probiotic Lozenge in the Treatment of Residual Pockets After Classical Non-surgical Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: s57667
Record Dates: First submitted 2015-05-06; First posted 2015-07-07 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Probiotic tablet
  Interventions: Other: Probiotic tablet- Biogaia
- Control (Placebo Comparator): Control tablet
  Interventions: Other: Placebo tablet

INTERVENTIONS:
Other: Probiotic tablet- Biogaia
  Arms: Test
Other: Placebo tablet
  Arms: Control

SUMMARY:
The aim of this study is to determine the efficacy of the usage of a probiobitc lozenge in patients with residual bleeding pockets of ≥ 5mm 3 months following scaling and rootplaning. Simultaneously the additional benefit of subgingival application of probiotics via oil drops will be investigated.

DETAILED DESCRIPTION:
The aim of this study is to determine the efficacy of the usage of a probiobitc lozenge in patients with residual bleeding pockets of ≥ 5mm following scaling and rootplaning. Simultaneously the additional benefit of subgingival application of probiotics via oil drops will be investigated.

Recruitment: This study will be a single centre (Department of Oral Health Sciences, University Hospitals Leuven), double blind, randomized, placebo controlled clinical trial with within each patient a split mouth design. The randomization (by means of a computer program) and double blind design are thought to minimize the bias of the investigator and patients.

Selection of the study population: Adults, who consult at the department of Periodontology at the University Hospital Leuven, and who fit the inclusion criteria will be asked to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* 40 patients
* ≥ 18 years of age
* scaling and rootplaning received at least 3 months ago
* Patients diagnosed with residual pockets (at least 2), with the definition of residual pockets:> 5mm or 5 and BOP+
* Willing and able to give written informed consent

Exclusion Criteria:

* patients with aggressive periodontitis
* patients who smoke
* pregnant or lactating woman
* patients with poorly controlled diabetes
* patients taking bisphosphonate mediation
* patient who had taken systemic antibiotics 3 months prior to treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Pocket Probing Depth (PPD) at teeth with residual pockets | 3-6 months
Recessions (REC) at teeth with residual pockets | 3-6 months
Clinical Attachment Loss (CAL) at teeth with residual pockets | 3-6 months

SECONDARY OUTCOMES:
Plaque at teeth with residual pockets | 3-6 months
Bleeding on Probing (BoP) at teeth with residual pockets | 3-6 months
Overall PPD, REC, CAL | 3-6 months
Microbial samples: deepest pocket, saliva, tongue | 3-6 months
Full Mouth Plaque Score (FMPS) and Full Mouth Bleeding Score (FMBS) | 3-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- UZLeuven, Leuven, Belgium